CLINICAL TRIAL: NCT04640155
Title: Treating Chronic Pouchitis With a Low FODMAP Diet
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study has been stopped due to difficulty with enrollment.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stephen Hanauer, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00213194
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Pouchitis
Keywords: Low FODMAP Diet; Pouchitis
MeSH Terms: conditions — Pouchitis | interventions — FODMAP Diet; Diet

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Diet (Other)
  Interventions: Behavioral: Regular Diet
- Low FODMAP (Experimental)
  Interventions: Behavioral: Low FODMAP Diet

INTERVENTIONS:
Behavioral: Low FODMAP Diet — Patients in the low FODMAP group will schedule a telephone visit with a registered dietician. During this approximately hour-long session, patients in the low FODMAP cohort will be counselled regarding FODMAP containing foods and how to effectively remove them while maintaining a nutrition-rich diet.
  Arms: Low FODMAP
Behavioral: Regular Diet — Patients in the regular diet group will receive an educational handout discussing low fiber diet, which is standard of care for those with pouchitis symptoms.
  Arms: Regular Diet

SUMMARY:
We aim to determine whether low FODMAP diet in patients with chronic pouchitis will improve symptoms and pouch inflammation.

DETAILED DESCRIPTION:
Following recruitment for entry into the study, subjects be asked to complete symptom surveys and provide a fecal sample for calprotectin measurement. Shortly after their screening visit, patients will be randomized 1:1 to either the low FODMAP diet (experimental) or regular diet (control) group. Patients in the experimental group will schedule a telephone visit with a registered dietician. During this approximately hour-long session, patients in the low FODMAP cohort will be counseled regarding FODMAP containing foods. They will be asked to adhere to this diet over the next 6 weeks. At the end of the 6 week period, subjects will complete a 3-day food diary. Those in the regular diet group will be contacted by the dietician and given an educational handout at the beginning of the study period regarding best dietary practices. At the end of the 6 week study period, both groups will again be asked to complete another set of symptom surveys and provide a fecal sample for calprotectin measurement.

ELIGIBILITY:
Inclusion Criteria

* Patients aged 18-65 with a diagnosis of ulcerative colitis that have undergone ileal pouch-anal anastomosis following proctocolectomy for medication-refractory disease
* Either ≥4 episodes of pouchitis per year (antibiotic-dependent) OR persistent symptoms despite 4 weeks of antibiotic therapy (antibiotic-resistant)

Exclusion Criteria

* Diagnosis of indeterminate colitis or Crohn's disease
* Celiac disease
* Current use of low FODMAP diet
* Known dietary allergies
* Current use of antibiotics for reasons other than treatment of pouchitis
* Clostridium difficile infection
* Complication following ileal pouch-anal anastomosis requiring reoperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Mean Difference in Fecal Calprotectin | 6 weeks

SECONDARY OUTCOMES:
Mean Difference in Composite Symptom Scores | 6 weeks
  Composite symptom score will include both clinical portion of Pouchitis Disease Activity Index as well as Oresland score, with possible scores ranging from 0-21 (higher number indicates higher symptom burden)
Mean Difference in Cleveland Global Quality of Life Score | 6 weeks
Rate of Normalization of Fecal Calprotectin | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Hanauer, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Medicine Digestive Health Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No